CLINICAL TRIAL: NCT00562263
Title: Barriers to Effective Weight Loss in Overweight Adolescents Enrolled in an Intensive, Team-based, Family-centered Lifestyle Modification Program
Brief Title: Barriers to Effective Weight Loss in Overweight Adolescents
Acronym: TEENS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HM11113
Record Dates: First submitted 2007-11-20; First posted 2007-11-22 (Estimated); Last update posted 2014-03-31 (Estimated); Status verified 2014-03

CONDITIONS: Overweight
Keywords: overweight; obesity; adolescent; insulin resistance; treatment
MeSH Terms: conditions — Overweight; Obesity; Insulin Resistance | interventions — Health

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lifestyle Modification (Experimental): Parents are randomized to attend 12 educational sessions covering strategies to manage children's health behaviors.
  Interventions: Behavioral: Lifestyle modification
- Control (No Intervention): Teen participates in lifestyle intervention, but parent does not attend parent education sessions

INTERVENTIONS:
Behavioral: Lifestyle modification — Dietary modification and regular physical activity
  Other Names: Weight Loss; Wellness
  Arms: Lifestyle Modification

SUMMARY:
The current study aims to investigate the impact of a comprehensive, team-based, family-centered, lifestyle modification program on body weight, metabolic abnormalities, fitness measures, and self-esteem in overweight adolescents beginning the study at ages 11-18 years. The intensive program will uniquely include a "team" structure and a component designed to address the role of parental modeling in effective lifestyle changes. By comparing the demographic, psychosocial, and metabolic characteristics of adolescents according to the degree of weight loss, the study will also more fully characterize the barriers that prevent successful participation in an intensive lifestyle modification program.

DETAILED DESCRIPTION:
The study will annually enroll 100 - 200 adolescent male and female subjects between 11 and 18 years of age with a BMI > the 85th percentile and one parent. Adolescents enrolled in the study, will participate in a structured exercise program and meet regularly with a dietitian and behavior specialist for nutrition education and review and update of progress and goals. The study is designed for 2 years of participation with data collection points at baseline, 3 months, 6 months, 1 year and 2 years. Data collected from adolescents include demographic information anthropometric information (height, weight, blood pressure, temperature, pulse, percent body fat); assessments of nutritional knowledge, food choices and dietary intake; assessments of activity and fitness level of behavioral status (depression, self-esteem, self-confidence, satisfaction with life, happiness, perspectives on health, exercise and diet, family environment, quality of life, body awareness, teasing, social efficacy, self-perception, coping mechanisms), assessments of sleep time and quality and physiological and medical data (including blood and urine tests)

Parents will accompany their children to the nutrition and behavior support visits, and attend 12 group educational sessions to learn skills and strategies to help their children adopt healthier eating and exercise behaviors. Data collected from parents will include demographic, anthropometric measures (height, weight, blood pressure, temperature, pulse, percent body fat); and assessments of activity level, dietary intake and eating habits, behavioral status, child-feeding practices, and understanding of their child.

ELIGIBILITY:
Inclusion Criteria:

* Age between 11 and 18
* BMI at or above the 85th percentile for age and sex
* At least one adult in the household who is committed to come to the program meetings

Exclusion Criteria:

* Previous enrollment in VCU IRB 3354
* Underlying genetic, neurologic, endocrine, or metabolic conditions that preclude weight loss with conventional diet and exercise programs
* Weight greater than 400 pounds
* Pregnancy in female adolescent subjects
* Inability to understand program instructions due to language barrier or a mental disability
* Primary residence outside a 30 mile radius program facility.
* Primary participating parent, if female, cannot be pregnant during the period corresponding to the parents intervention.

Ages: 11 Years to 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 257 (Actual)
Dates: Start 2007-10; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
changes in BMI Z-score | 3 month, 6 month, 12 months and 24 months

SECONDARY OUTCOMES:
Changes in body composition, metabolic and anthropometric measures, fitness measures, dietary intake, and quality of life scores. | 3 month, 6 month, 1 year and 2 years.

CONTACTS AND LOCATIONS:
Overall Officials: Gary L. Francis, M.D., Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

REFERENCES:
- [Derived] Ning Y, Yang S, Evans RK, Stern M, Sun S, Francis GL, Wickham EP 3rd. Changes in body anthropometry and composition in obese adolescents in a lifestyle intervention program. Eur J Nutr. 2014 Jun;53(4):1093-102. doi: 10.1007/s00394-013-0612-9. Epub 2013 Nov 10. PMID 24212451